CLINICAL TRIAL: NCT06819358
Title: Individualized Functional Imaging-Guided Repetitive Transcranial Magnetic Stimulation (rTMS) for Treating Postural Gait Disorders in Patients with Amyotrophic Lateral Sclerosis (ALS): a Randomized, Crossover, Controlled, Double-Blind Clinical Study
Acronym: iFIRST-ALS
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Changping Laboratory (Other)
Responsible Party: Principal Investigator, He Ji, Associate professor/Associate chief physician, Peking University Third Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M2024877
Record Dates: First submitted 2025-01-23; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: Individualized cortical mapping technology, repetitive transcranial magnetic stimulation, amyotrophic lateral sclerosis, balance and gait disorders.
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Mobility Limitation | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: This study is a randomized, crossover, controlled, double-blind clinical trial. Patients (n=45) were randomly divided into Group A and Group B. Patients in Group A will receive 2 weeks (10800 Hz daily, 5 days×2) of TMS treatment, while patients in Group B will receive sham stimulation with the same frequency. After a 4-week washout period, the two groups cross over. Patients in Group A will receive sham stimulation, and patients in Group B will receive TMS treatment for 2 weeks (10800 Hz daily, 5 days×2). Clinical functional scales, imaging evaluations, and gait analysis will be conducted at baseline, after 2 weeks of treatment, before crossover treatment, and after 2 weeks of crossover treatment. The therapist, patients, and assessors will be all blinded throughout the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator)
  Interventions: Device: Transcranial Magnetic Stimulation
- Group B (Sham Comparator)
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Patients in Group A will receive 2 weeks (10800 Hz daily, 5 days×2) of TMS treatment, while patients in Group B will receive sham stimulation with the same frequency. After a 4-week washout period, the two groups cross over. Patients in Group A will receive sham stimulation, and patients in Group B will receive TMS treatment for 2 weeks (10800 Hz daily, 5 days×2).

SUMMARY:
This study is a randomized, crossover, controlled, double-blind clinical trial. Patients (n=45) were randomly divided into Group A and Group B. Patients in Group A will receive 2 weeks (10800 Hz daily, 5 days×2) of Transcranial magnetic stimulation（TMS） treatment, while patients in Group B will receive sham stimulation with the same frequency. After a 4-week washout period, the two groups cross over. Patients in Group A will receive sham stimulation, and patients in Group B will receive TMS treatment for 2 weeks (10800 Hz daily, 5 days×2). Clinical functional scales, imaging evaluations, and gait analysis will be conducted at baseline, after 2 weeks of treatment, before crossover treatment, and after 2 weeks of crossover treatment. The therapist, patients, and assessors will be all blinded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-80 years;
2. Diagnosis of motor neuron disease at probable level or above based on Estorial criteria;12
3. Meet UMND ALS diagnosis criteria: at least three segments of upper motor neuron damage localized to 1-2 muscles, or EMG indicating loss of innervation in 1-2 muscles;13
4. Presence of lower limb dysfunction: Berg balance scale score below 40;
5. Capable of standing independently for more than 30 seconds and able to walk or walk with assistance;
6. Stable medication dosage for at least one month;
7. FVC > 60%;
8. Signed informed consent.

Exclusion Criteria:

1. History of substance abuse within the past 6 months;
2. History of epilepsy or first-degree relative with epilepsy;
3. Patients with severe systemic diseases in the heart, lungs, liver, or kidneys that cannot be controlled with routine medications, based on laboratory results;
4. Patients with severe depression or anxiety (HAMD-17 score ≥18; HAMA score ≥21) or diagnosed with other mental illnesses;
5. Patients with a life expectancy of less than one year due to reasons other than neurodegenerative diseases;
6. Pregnant women or those planning to become pregnant;
7. Individuals with a pacemaker, cochlear implant, or other metallic foreign bodies and any implanted electronic equipment, or those with contraindications for MRI scanning or TMS treatment, such as claustrophobia;
8. Patients who have received TMS, transcranial electrical stimulation, transcranial focused ultrasound, or other neuromodulation treatments within three months prior to enrollment;
9. Other abnormal examination results deemed unsuitable for participation by the research investigator;
10. Inability to cooperate for follow-ups due to geographical or other reasons;
11. Participation in other clinical research trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-02-14 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Scale evaluation | Baseline (Week 0), Week 2, Week 6, Week 8
  The Berg Balance Scale (BBS) assesses static and dynamic balance. The scale ranges from 0 to 56, with higher scores indicating better balance and lower scores signifying greater fall risk.

SECONDARY OUTCOMES:
Scale evaluation | Baseline (Week 0), Week 2, Week 6, Week 8
  Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) Total Score(ALSFRS-R total score).The ALSFRS-R evaluates functional impairment in ALS patients. The total score ranges from 0 to 48, with higher scores reflecting better functional ability.
Scale evaluation | Baseline (Week 0), Week 2, Week 6, Week 8
  Walking and stepping sub-items, Modified Ashworth Scale (MAS),The scale ranges from 0 to 4, with higher scores indicating greater spasticity.
Scale evaluation | Baseline (Week 0), Week 2, Week 6, Week 8
  Timed Instant Walking (TUG) tes,the TUG test measures mobility and fall risk. Lower times indicate better mobility.
Scale evaluation | Baseline (Week 0), Week 2, Week 6, Week 8
  10-meter walking test time (10MWT),This test measures walking speed over a 10-meter distance. Lower times indicate faster walking speed
Imaging evaluation | Baseline (Week 0), Week 2, Week 6, Week 8
  Functional MRI (fMRI) - Brain Function and Cortical Excitatory Changes, fMRI will assess changes in brain function and cortical excitability.Functional MRI (fMRI) is a neuroimaging technique used to assess brain function by detecting changes in blood oxygen levels (BOLD signal), which reflect neural activity. In this study, fMRI will be used to evaluate brain function and cortical excitability in patients with schizophrenia. Specifically, it will assess neural activation patterns in response to cognitive and emotional tasks designed to probe social cognition, emotion recognition, and executive functions. Areas of interest include the prefrontal cortex, amygdala, and visual processing regions involved in emotion processing and decision-making.fMRI will be performed as follows:Participants will be scanned while completing emotion recognition tasks to identify brain regions activated during these tasks.Scans will be conducted in a resting-state condition as well, to measure baseline cort
Gait instrument | Baseline (Week 0), Week 2, Week 6, Week 8
  Gait Assessment and Fall Index (Tetrax Instrument),Gait and fall risk assessment will be conducted using the Tetrax instrument. Data will be analyzed as index. The Fall Index Assessment is conducted using the Tetrax instrument, which is a widely used device for evaluating balance and fall risk. The Tetrax system consists of a set of sensors placed on the patient's feet to measure their ability to maintain balance in various postural positions, including static (standing still) and dynamic (movement) tasks. The system evaluates several components of balance, including:Postural Sway: The extent of body movement while standing;Stability: The ability to maintain a balanced posture under different conditions;Response Time: How quickly the subject can correct their posture after perturbation (e.g., slight push)；Foot Pressure Distribution: How evenly weight is distributed between the feet while standing.
biological indicator | Baseline (Week 0), Week 2, Week 6, Week 8
  Neurofilament protein (NFL),NFL levels will be measured in blood samples to assess neurodegeneration.Neurofilament light chain (NFL) is measured in peripheral blood samples using the SIMOA (Single Molecule Array) assay, a highly sensitive technique that quantifies NFL levels at the single-molecule level. NFL concentration is expressed in pg/mL, with higher levels indicating greater neuronal injury or neurodegeneration.

IPD SHARING:
Plan to Share IPD: Undecided